CLINICAL TRIAL: NCT06993675
Title: Improving MRD Negativity Rates in Newly Diagnosed Multiple Myeloma Patients: a Response-adaptive Approach of Consolidation With One or Two Bispecific T-cell Engagers Against GPRC5D or BCMA
Brief Title: Engaging T-cells to Eliminate MRD in Newly Diagnosed Myeloma Optimizing Response With Talquetmab and Teclistamab (ROTATE)
Acronym: ROTATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Noffar Bar (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Noffar Bar, Assistant Professor of Medicine (Hematology), Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000038510
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: minimal residual disease; ROTATE
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Talquetamab is a GPRC5DxCD3 bispecific antibody. It is supplied as a sterile, preservative-free solution for subcutaneous administration.
  Teclistamab is a BCMAxCD3 bispecific antibody. It is supplied as a sterile, preservative-free solution for subcutaneous administration.
  Interventions: Drug: Talquetamab; Drug: Teclistamab

INTERVENTIONS:
Drug: Talquetamab — Talquetamab is a GPRC5DxCD3 bispecific antibody. It is supplied as a sterile, preservative-free solution for subcutaneous administration.
Drug: Teclistamab — Teclistamab is a BCMAxCD3 bispecific antibody. It is supplied as a sterile, preservative-free solution for subcutaneous administration.

SUMMARY:
Multiple myeloma is characterized by a pattern of recurrent relapse and remains an incurable malignancy. Participants with minimal residual disease (MRD) after front line therapy with induction with or without transplant have worse prognosis than those with MRD negative disease.

Bispecific T-cell-based immunotherapies have the potential to promote further reduction of malignant plasma cells thus improving rates of MRD negativity and improve patient outcomes. In this study, participants who are MRD positive after front line therapy will receive consolidation with GPRC5D-targeted bispecific talquetamab. We will test MRD negative conversion and if MRD negativity was not achieved, the participant will switch to a different target using the B-cell maturation antigen TCE, teclistamab. Consolidation will be continued for up to 1 year in participants who have achieved MRD negativity.

ELIGIBILITY:
Inclusion Criteria

To qualify for participation in this study, an individual must satisfy each of the following criteria:

1. Provision of signed and dated ICF.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female aged 18 years or older.
4. Newly diagnosed multiple myeloma participants who are transplant eligible and have completed at least four cycles of quadruplet, anti-CD38 antibody-based induction and have received HDM ASCT within 60-120 days. If consolidation with the same induction regimen is used post ASCT, enrolment up to 60 days post consolidation.
5. Must have MRD positive disease at 10-5 based on NGS with a PR or better response.
6. Must not be progressing as per IMWG criteria
7. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale of 0 or 1. ECOG 2 or 3 are eligible for the study if the ECOG PS score is related to stable physical limitations (e.g., wheelchair-bound due to prior spinal cord injury) and not related to multiple myeloma or associated therapy. Adequate bone marrow function:

   1. Hemoglobin 8 g/dl (³5mmol/L; without prior RBC transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted).
   2. Absolute neutrophil count ≥1.0×109/L (prior growth factor support is permitted but must be without support for 7 days for G-CSF or GM-CSF and for 14 days for pegylated-G-CSF).
   3. Platelets ³75×109/L (without transfusion support or thrombopoietin receptor agonist within 7 days before the laboratory test).
8. Estimated creatinine clearance ≥30 mL/min based on the Cockcroft-Gault Equation (see https://www.mdcalc.com/calc/43/creatinine-clearance-cockcroft-gault-equation)
9. Must have adequate liver function:

   1. Aspartate aminotransferase ≤2.5 folds of the upper limit of normal (ULN).
   2. Alanine aminotransferase ≤2.5 folds of the ULN.
   3. Serum bilirubin ≤ 1.5 x ULN (except in participants with congenital bilirubinemia, such as Gilbert syndrome where must be <5xULN).
10. Participants must adhere to the following reproductive and contraceptive requirements while on study treatment and for the specified duration after the last dose of talquetamab or teclistamab:

    1. For participants receiving talquetamab, these criteria apply for three months after the last dose.
    2. For participants receiving teclistamab, these criteria apply for five months for those assigned female at birth and three months for those assigned male at birth.
    3. General Requirements:

    i. Participants must not be pregnant or breastfeeding. ii. Participants must not donate gametes (i.e., eggs or sperm) or freeze gametes for future use related to assisted reproduction.

    d. For participants of childbearing potential: Participant of childbearing potential is defined as an individual who is premenopausal and capable of becoming pregnant, including those using contraception, those who are single, or those with partners who have had a vasectomy.

ii. A negative highly sensitive pregnancy test must be obtained at screening within 24 hours before the first dose of talquetamab (first study treatment), and participants must agree to further pregnancy tests throughout the study.

iii. Participants must practice at least one highly effective method of contraception.

e. For Partners of Participants: i. If the participant's partner is of childbearing potential, the partner must also practice a highly effective method of contraception while the participant is on study treatment and for three months after the last dose of talquetamab or the last dose of teclistamab, unless the participant is vasectomized.

f. Highly effective methods of contraception include, but are not limited to: i. Combined hormonal contraception (estrogen and progestogen) that inhibits ovulation (oral, intravaginal, or transdermal).

ii. Progestogen-only hormonal contraception that inhibits ovulation (oral, injectable, or implantable).

iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system. v. Bilateral tubal occlusion. vi. Sexual abstinence (the reliability of abstinence must be evaluated concerning the duration of the clinical study and the participant's lifestyle).

vii. A vasectomized partner (provided the partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has received medical confirmation of the surgical success).

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Prior or concurrent exposure to any of the following within the specified timeframe prior to randomization:

   1. Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or ≥5 half-lives, whichever is less.
   2. Investigational vaccine within four weeks.
   3. Monoclonal antibody therapy within 21 days.
   4. Cytotoxic therapy within 14 days.
   5. PI therapy within 14 days.
   6. IMiD agent therapy within 14 days.
   7. Radiotherapy within 14 days or focal radiation within seven days.
   8. Gene-modified adoptive cell therapy (e.g., chimeric antigen receptor modified T-cells, NK cells) within three months.
   9. Prior exposure to a bispecific T-cell engager or CAR T-cell therapy.
2. An active or suspected infection at time of screening. For rescreening refer to section 5.5.
3. Known history or serologic evidence of human immunodeficiency virus (HIV) infection.
4. Known history, virologic, or serological evidence of hepatitis B or C virus (HBV/HCV) infection; participants who had HCV but have received an antiviral treatment and show no detectable HCV viral RNA for six months are eligible. Participants with no active hepatitis B infection (e.g., HBsAg negative, anti-HBcAb positive) who are under adequate prophylaxis per local standard of care against HBV reactivation may be eligible.
5. Class III or IV congestive heart failure.
6. Presence of clinically relevant CNS pathology.
7. Another active malignancy that requires treatment.
8. Pregnancy or lactation.
9. Known allergic reactions to components of talquetamab or teclistamab.
10. Received a cumulative dose of corticosteroids equivalent to ≥140 mg of prednisone within 14 days before first dose of study drug.
11. Received a live, attenuated vaccine within four weeks before the first dose of study drug.
12. Plasma cell leukemia, smoldering multiple myeloma, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary light chain amyloidosis.
13. Any active malignancy (i.e., progressing or requiring treatment change in the last 24 months) other than multiple myeloma. The only allowed exceptions are malignancies treated within the last 24 months that are considered cured:

    1. Non-muscle invasive bladder cancer (solitary Ta-PUN-LMP or low grade, <3 cm, no CIS).
    2. Non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone.
    3. Non-invasive cervical cancer.
    4. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ or history of localized breast cancer (anti-antihormonal therapy is permitted).
    5. Localized prostate cancer (M0, N0) with a Gleason Score ≤7a, treated locally only (RP/RT/focal treatment).
    6. Other malignancy that is considered cured with minimal risk of recurrence in consultation with the sponsor-investigator.

    NOTE: In the event of any questions, consult with the sponsor-investigator prior to enrolling a participant.
14. Stroke, transient ischemic attack or seizure within six months prior to enrolment.
15. Presence of the following cardiac conditions:

    1. New York Heart Association stage III or IV congestive heart failure (Appendix 5: New York Heart Association Functional Classification).
    2. Myocardial infarction, unstable angina, or coronary artery bypass graft ≤6 months prior to randomization.
    3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.
    4. Uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities.
16. Major surgery within two weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within two weeks after administration of the last dose of study treatment.

    NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a participant in the study.
17. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

    1. Acute diffuse infiltrative pulmonary disease
    2. Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy
    3. Active autoimmune disease requiring systemic immunosuppressive therapy within six months before start of study treatment. Exception: Participants with vitiligo, controlled type I diabetes, and prior autoimmune thyroid disease that is currently euthyroid based on clinical symptoms and laboratory testing are eligible regardless of when these conditions were diagnosed.
    4. Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status
    5. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
    6. History of noncompliance with recommended medical treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD Negative Response at 10^-5 Sensitivity Using NGS ClonoSEQ Assay in Participants with Newly Diagnosed Multiple Myeloma Treated with Talquetamab Consolidation With or Without Sequential Teclistamab by 12 Months | 12 months from the start of treatment
  The primary outcome measure will evaluate the efficacy of talquetamab consolidation therapy, with or without the sequential use of teclistamab, by assessing the rate of minimal residual disease (MRD) negative response at a sensitivity level of 10^-5. This evaluation will be conducted using the next-generation sequencing (NGS) ClonoSEQ assay. The primary endpoint is the proportion of participants who achieve MRD negativity at 10^-5 sensitivity after consolidation therapy with talquetamab, with or without the sequential use of teclistamab, by 12 months from the start of treatment. MRD negative response is defined as the absence of detectable myeloma cells in bone marrow, as determined by the highly sensitive NGS ClonoSEQ assay. This measure aims to determine the depth of response and the potential of the treatment regimen to achieve sustained deep remission in participants with newly diagnosed multiple myeloma.

SECONDARY OUTCOMES:
Complete Response and MRD-Negative Complete Response in Multiple Myeloma Patients Treated with Talquetamab Consolidation, With or Without Sequential Teclistamab | At baseline then at Cycle 7, each cycle is 28 days
  To evaluate the achievement of complete response (CR) or better, including MRD-negative complete response, in patients with multiple myeloma who are treated with talquetamab as a consolidation therapy. The assessment will include both scenarios: talquetamab used alone and talquetamab followed by sequential teclistamab. This evaluation aims to provide insights into the depth of response and eradication of minimal residual disease in the treated cohorts.
Assessment of Minimal Residual Disease (MRD) at 10^-6 Sensitivity in Multiple Myeloma Patients | At baseline then at Cycle 7, each cycle is 28 days
  To assess the level of minimal residual disease (MRD) at a sensitivity threshold of 10^-6 in patients with multiple myeloma undergoing treatment. This high sensitivity assessment aims to determine the extent of disease eradication and to provide a deeper understanding of the effectiveness of the therapeutic regimen in achieving nearly undetectable levels of remaining cancer cells.
Determination of Sustained MRD-Negative Rate at One Year in Multiple Myeloma Patients | One year post-treatment
  To determine the sustained minimal residual disease (MRD) negative rate one year post-treatment in patients with multiple myeloma. This measure aims to evaluate the durability of the MRD-negative status over a one-year period, providing insights into the long-term efficacy of the treatment regimen in maintaining deep and persistent disease remission.
Quality of Life Assessment via Patient-Reported Outcomes in Response to Treatment | Day 1 of Cycles 1-6, where each cycle is 28 days, then at EOT(treatment durations is 15-24 months) and Safety Follow-Up visits(patients will be followed for 6 months)
  To evaluate the quality of life (QoL) of patients with multiple myeloma through patient-reported outcome measures in response to the treatment regimen. This assessment aims to capture the subjective experiences of patients, including physical, emotional, and social well-being, to gain a comprehensive understanding of how the treatment impacts their overall quality of life. Patient-reported outcomes will provide valuable insights into the effectiveness of the therapy from the perspective of those undergoing treatment.
Assessment of Treatment-Related Adverse Events in Multiple Myeloma Patients | From baseline till the first safety follow-up visit; approximately 15-24 months
  To assess the incidence and severity of treatment-related adverse events in patients with multiple myeloma undergoing the specified therapeutic regimen. This evaluation aims to systematically document and analyze any negative side effects or complications associated with the treatment, providing crucial safety data and helping to weigh the risks against the potential benefits of the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Noffar Bar, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No